CLINICAL TRIAL: NCT00287339
Title: Chronic Cough and Reflux Disease: A Randomized, Double-Blinded, Placebo Controlled Trial of High Dose Proton Pump Inhibition
Brief Title: The Utility of Nexium in Chronic Cough and Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Nicholas Shaheen, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ COUGH
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Cough; GERD
Keywords: Cough; GERD
MeSH Terms: conditions — Cough; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 40mg Esomeprazole BID
  Interventions: Drug: Esomeprazole
- 2 (Placebo Comparator): placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 40mg capsule BID for 12 weeks
  Other Names: Brand name is Nexium
  Arms: 1
Drug: Placebo — placebo capsule BID for 12 weeks
  Arms: 2

SUMMARY:
The purpose of this research study is to investigate different doses of proton pump inhibitors in reducing cough symptoms felt to be associated with Gastroesophageal reflux disease (GERD). Proton pump inhibitors are medicines used to treat GERD, which work by lowering the amount of acid in the stomach.

The proton pump inhibitor used in this study is called, Esomeprazole (brand name Nexium), and is already marketed for treating GERD. Patients with GERD may experience all or some of the following symptoms: stomach acid or partially digested food re-entering the esophagus (which is sometimes referred to as heartburn or regurgitation), belching and coughing. Even very small, unnoticeable amounts of rising stomach acid may cause patients to cough.

Because there may be a link between chronic cough and GERD, study doctors are interested in learning if giving high-dose Nexium (40 milligrams, twice daily) will help in treating chronic cough.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo controlled, comparative parallel-group trial of subjects with chronic cough of unknown origin presenting to the Otolaryngology/ Head and Neck Surgery, Pulmonary Medicine, and Gastroenterology outpatient clinics at the University of North Carolina Hospital system.

Potential subjects with chronic cough of unknown origin will be identified through the above outpatient clinics. Those who meet the inclusion and exclusion criteria will be asked to join the study testing the efficacy of twice daily esomeprazole 40 mg taken for 3 months in the setting of chronic cough. Potential subjects will be consented for the study prior to leaving the enrolling clinic. A total of 40 subjects will be recruited into our study.

ELIGIBILITY:
Inclusion Criteria:

1. males and females (of non-childbearing potential. ie-surgically sterile, or willing to use an approved form of birth control) between the ages of 18 and 70 who speak and write in English,
2. chronic cough (> 8 wks/another article used > 6 wks) with symptom severity criteria of 2 or greater on the Fisman Cough Severity Score and 3 or greater or the Fisman Cough Frequency Score, and,
3. failure to respond to post nasal drip therapy.

Exclusion Criteria:

1. abnormal chest x-ray,
2. patients taking H2 blockers within the previous 3 days or PPI's within the previous 7 days,
3. failure to respond to past PPI therapy given for cough that lasted at least 12 weeks,
4. use of an investigational drug within the past 30 days,
5. previous surgical antireflux or non-surgical endoscopic anti-reflux procedure (ex., Stretta or endoscopic sewing device),
6. previous aerodigestive malignancy,
7. current smokers, or ex-smokers (defined as those who quit smoking less than 3 months prior to study enrollment or those who have quit, but have a 20 pack year smoking history),
8. upper respiratory infection within 8 weeks prior to study enrollment,
9. current use of a B- blocker, ACE-I, or anticholinesterases at time of enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Gastroenterology
Locations (1):
- UNC Gastroenterology, UNC Pulmonology, UNC ENT, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Shaheen NJ, Crockett SD, Bright SD, Madanick RD, Buckmire R, Couch M, Dellon ES, Galanko JA, Sharpless G, Morgan DR, Spacek MB, Heidt-Davis P, Henke D. Randomised clinical trial: high-dose acid suppression for chronic cough - a double-blind, placebo-controlled study. Aliment Pharmacol Ther. 2011 Jan;33(2):225-34. doi: 10.1111/j.1365-2036.2010.04511.x. Epub 2010 Nov 17. PMID 21083673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited from hospital clinics - subjects with chronic cough.
Pre-assignment Details: . After initial eligibility screening, all consenting participants entered a 7-day run-in period, during which all subjects took a placebo pill twice a day, for the purpose of ensuring compliance with study medication and assessment of cough severity under baseline conditions.
Groups:
- Esomeprazole Arm: Upon successful completion of the run-in period, participants in the esomeprazole arm were given the compound at a dose of 40mg for 12 weeks. All participants were instructed to take their study medication 30 minutes before breakfast and 30 minutes before dinner. Esomeprazole was supplied by the investigational pharmacy at the University of North Carolina as blue capsules without identifying features.
- Placebo: Upon successful completion of the run-in period, participants randomized to receive to the placebo arm got a capsule identical to the esomeprazole arm, but containing an inert substance, twice daily for 12 weeks. All participants were instructed to take their study medication 30 minutes before breakfast and 30 minutes before dinner.
Period: Overall Study
Arm/Group | Esomeprazole Arm | Placebo
Started | 22 | 18
Completed | 22 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole Arm | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12) | 51.0 (11.6) | 50 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough-Specific Quality of Life Questionnaire
Description: It is a validated, 28-item assessment tool designed to evaluate decrements in quality of life due to chronic cough. This questionnaire measures cough-related symptoms, as well as the social implications and psychological impact. Examples of items include, "I cannot sleep at night" and "I cough and it makes me retch." The final score is obtained by summing the responses to 28 questions, each scored on a 1-4 scale, where 1 is "strongly disagree," and 4 is "strongly agree." The minimum and maximum CQLQ scores are 28 and 112 respectively, with increasing score indicating more severe impairment.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Esomeprazole Arm | Placebo
Number analyzed (Participants) | 22 | 18
participants | 9.8 (12.2) | 5.8 (11.1)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Esomeprazole Arm | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

LIMITATIONS AND CAVEATS:
This study was performed at a single center, and participants were mostly female and white, which may limit generalizability. The number of subjects in some patient subgroups was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No